CLINICAL TRIAL: NCT05880407
Title: Pilot Study of Percutaneous Correction of Hallux Valgus: Clinical-functional Evaluation of Outcome Randomized Study
Brief Title: Pilot Study of Percutaneous Correction of Hallux Valgus
Acronym: hallux valgus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hallux valgus
Record Dates: First submitted 2023-02-01; First posted 2023-05-30 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment (Active Comparator): SERI osteotomy
  Interventions: Procedure: SERI osteotomy
- experimental treatment (Experimental): percutaneous osteotomy according to Chevron
  Interventions: Procedure: percutaneous osteotomy according to Chevron

INTERVENTIONS:
Procedure: SERI osteotomy — Correction of varus deformity of the 1st Metatarsal that is stabilized with Kirschnner wire
  Arms: standard treatment
Procedure: percutaneous osteotomy according to Chevron — Correction of varus deformity by osteotomy stabilization with 2 screws inserted via dorsal percutaneous accesses to the 1st Metatarsal.
  Arms: experimental treatment

SUMMARY:
This is a pilot study with a randomized controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with adult hallux valgus with indication for corrective surgical treatment
* HVA (hallux valgus angle): 20°-40°
* IMA (intermetatarsal angle): 10°-20°

Exclusion Criteria:

* Patients with instability of the first metatarsophalangeal joint
* Patients with severe morphostructural alterations or other pathologies in the foot and lower limb
* patients requiring additional surgical procedures
* patients with severe vascular and neurological systemic pathologies
* systemic pathologies that may impair bone consolidation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score | baseline
  pain visual analog assessment
Visual Analog Score | 1 year
  pain visual analog assessment

SECONDARY OUTCOMES:
American Orhtopaedic Foot and Ankle Society forefoot score | baseline and aftef 1 year
  range of motion evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy